CLINICAL TRIAL: NCT05818904
Title: Ultrasound Imaging of Fibrotic Tissue Using Machine Learning
Brief Title: Ultrasound Imaging of Fibrotic Tissue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhou Mouwang, Professor, Peking University Third Hospital
Other Study IDs: M2022793
Record Dates: First submitted 2023-03-08; First posted 2023-04-19 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Arthrofibrosis of Knee; Arthrofibrosis of Shoulder
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: Healthy group is recruited. They would not receive any intervention. The ultrasound imaging data will be collected to serve as the comparison for no fibrosis joint.
- Arthrosis of knee: People with arthrosis of the knee joint will be treated using the traditional intervention, which includes physical therapy. The ultrasound imaging will be collected before the intervention and at 3-month. The imaging data will be used to build a imaging model using the machine learning method.
  Interventions: Other: Physical Therapy
- arthrosis of shoulder: People with arthrosis of the shoulder joint will be treated using the traditional intervention, which includes physical therapy. The ultrasound imaging will be collected before the intervention and at 3-month. The imaging data will be used to build a imaging model using the machine learning method.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — All arthrosis participants will be treated as the traditional methods using physical therapy.
  Groups: Arthrosis of knee; arthrosis of shoulder

SUMMARY:
This project intends to collect the ultrasonic spectrum information of shoulder and knee joint fibrotic tissue, and use machine learning to study the mechanism of fibrosis tissue ultrasound imaging, and then build a model and finally establish the relationship between joint stiffness and fibrosis formation. In this study, the broadband ultrasound imaging method for joint fibrosis has the potential to create a method for ultrasonic localization, staining and evaluation of joint fibrosis, laying the foundation for the research of new conservative treatment methods and surgical positioning for fibrosis, and for reducing the occurrence of joint fibrosis rate, improve joint function of patients, and return to family and society earlier and better

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral shoulder or knee joint stiffness and normal on the opposite side
2. The course of the disease is longer than 3 months
3. Good cognitive function, able to understand the content of this experiment, willing to cooperate with follow-up
4. Over 18 years old, voluntarily participate in this study, and sign the informed consent

Exclusion Criteria:

1. Wound non-healing, joint dislocation or unstable fracture fixation, pseudarthrosis, joint purulent infection and other contraindications for joint range of motion examination
2. There are skin lesions, wounds or allergies to the coupling agent on the joint surface and other conditions that cannot be used for ultrasound examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Joint stiffness patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
KOOS score | 3-month
  The KOOS (Knee injury and Osteoarthritis Outcome Score) survey is a health questionnaire used to assess the impact of knee injury or osteoarthritis on patients. It has 42 questions covering 5 domains and is rated on a 5-point Likert scale. The scale ranges from 0 to 100, with higher scores indicating better outcomes. The KOOS survey is a reliable and valid tool used in research and clinical practice to assess treatment effectiveness and track symptom changes over time.
CM score | 3-month
  The Constant-Murley survey is a health questionnaire used to evaluate shoulder function and pain. It consists of four domains: pain, activities of daily living, range of motion, and strength. The scale ranges from 0 to 100, with higher scores indicating better outcomes. The Constant-Murley survey is a reliable and valid tool used in research and clinical practice to assess treatment effectiveness and track symptom changes over time.

SECONDARY OUTCOMES:
SF-36 | 3-month
  The SF-36 (36-Item Short Form Survey) is a health questionnaire used to measure general health and well-being. It consists of 36 questions that evaluate eight domains, including physical functioning, role limitations, pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. The scale ranges from 0 to 100, with higher scores indicating better outcomes. The SF-36 survey is a widely used and reliable tool used in research and clinical practice to assess health status and well-being.
WOMAC | 3-month
  The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) survey is a health questionnaire used to evaluate the severity of osteoarthritis in the knee and hip joints. It consists of 24 questions that evaluate three domains, including pain, stiffness, and physical function. The scale ranges from 0 to 96, with higher scores indicating worse outcomes. The WOMAC survey is a reliable and valid tool used in research and clinical practice to assess treatment effectiveness and track symptom changes over time.
HSS-KS | 3-month
  The HSS (Hospital for Special Surgery) survey is a health questionnaire used to assess patient outcomes after total hip or knee replacement surgery. It consists of 40 questions that evaluate patient pain, function, and satisfaction with the surgery. The scale ranges from 0 to 100, with higher scores indicating better outcomes. The HSS survey is a reliable and valid tool used in research and clinical practice to assess treatment effectiveness and track patient satisfaction and function over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No